CLINICAL TRIAL: NCT01009593
Title: An Open-label, Randomized Phase 3 Study of the Efficacy and Tolerability of Linifanib (ABT-869) Versus Sorafenib in Subjects With Advanced Hepatocellular Carcinoma (HCC)
Brief Title: Efficacy and Tolerability of ABT-869 Versus Sorafenib in Advanced Hepatocellular Carcinoma (HCC)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M10-963; 2009-013435-38 (EudraCT Number)
Record Dates: First submitted 2009-10-14; First posted 2009-11-06 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-06

CONDITIONS: Hepatocellular Carcinoma Non-resectable; Hepatocellular Carcinoma Recurrent; Carcinoma, Hepatocellular; Liver Diseases; Neoplasms by Histologic Type; Digestive System Neoplasms; Carcinoma; Liver Neoplasms; Neoplasms; Neoplasms by Site; Digestive System Diseases; Adenocarcinoma; Neoplasms, Glandular and Epithelial
Keywords: Molecular Mechanisms of Pharmacological Action; Antineoplastic Agents; Growth Substances; Physiological Effects of Drugs; Enzyme Inhibitors; Angiogenesis Inhibitors; Inhibitors, Angiogenesis; Protein Kinase Inhibitors; Pharmacologic Actions; Growth Inhibitors; Angiogenesis Modulating Agents; Sorafenib
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Diseases; Neoplasms by Histologic Type; Digestive System Neoplasms; Carcinoma; Liver Neoplasms; Neoplasms; Neoplasms by Site; Digestive System Diseases; Adenocarcinoma; Neoplasms, Glandular and Epithelial | interventions — linifanib; Sorafenib

ARMS (2):
- ABT-869 (Experimental)
  Interventions: Drug: ABT-869
- Sorafenib (Active Comparator)
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: ABT-869 — Tablets, Oral, 17.5 mg, Once Daily, Until disease progression or unacceptable toxicity
  Arms: ABT-869
Drug: Sorafenib — Tablets, Oral, 400 mg, Twice Daily, Until disease progression or unacceptable toxicity.
  Arms: Sorafenib

SUMMARY:
The primary objective of this study is to assess the overall survival (OS) of oral linifanib given as monotherapy once daily (QD) compared to sorafenib given twice daily (BID) per standard of care in subjects with advanced or metastatic HCC.

DETAILED DESCRIPTION:
The IDMC recommended discontinuation of the study, and, the protocol was amended to end study treatment.

ELIGIBILITY:
Inclusion Criteria

* Histologic or cytologic diagnosis with unresectable or metastatic HCC
* Child Pugh Class A
* ECOG performance status 0-1
* Adequate hematologic, hepatic, and renal function

Exclusion Criteria

* Prior systemic (administered intravenously or orally rather than locoregionally) treatment for HCC
* Prior local therapy (including liver-directed therapy) within 4 weeks from entry
* Untreated brain or meningeal metastases
* Current treatment on another clinical trial
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1035 (Actual)
Dates: Start 2010-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Overall Survival | From randomization until patient death; assessed monthly

SECONDARY OUTCOMES:
Time To Progression (TTP) | From randomization until patient progression; assessed every 6 weeks
Overall Response Rate (ORR) | Assessed Every 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Justin Ricker, MD, Study Director — Abbott
Locations (163):
- United States (13):
  - Site Reference ID/Investigator# 23247, Beverly Hills, California
  - Site Reference ID/Investigator# 23608, LaVerne, California
  - Site Reference ID/Investigator# 23852, Orange, California
  - Site Reference ID/Investigator# 40162, Orange, California
  - Site Reference ID/Investigator# 23254, Newark, Delaware
  - Site Reference ID/Investigator# 23253, Gainesville, Georgia
  - Site Reference ID/Investigator# 23609, Honolulu, Hawaii
  - Site Reference ID/Investigator# 24848, Honolulu, Hawaii
  - Site Reference ID/Investigator# 23250, Louisville, Kentucky
  - Site Reference ID/Investigator# 23257, St Louis, Missouri
  - Site Reference ID/Investigator# 23603, Las Vegas, Nevada
  - Site Reference ID/Investigator# 23244, Durham, North Carolina
  - Site Reference ID/Investigator# 23252, Portland, Oregon
- Argentina (2):
  - Site Reference ID/Investigator# 35705, Buenos Aires
  - Site Reference ID/Investigator# 35702, Rosario, Santa Fe
- Australia (5):
  - Site Reference ID/Investigator# 23152, Camperdown
  - Site Reference ID/Investigator# 23150, Concord
  - Site Reference ID/Investigator# 27122, Kingswood
  - Site Reference ID/Investigator# 23153, Kogarah
  - Site Reference ID/Investigator# 24103, Southport
- Austria (4):
  - Site Reference ID/Investigator# 27968, Graz
  - Site Reference ID/Investigator# 27969, Innsbruck
  - Site Reference ID/Investigator# 27970, Linz
  - Site Reference ID/Investigator# 27967, Vienna
- Belgium (6):
  - Site Reference ID/Investigator# 38902, Brussels
  - Site Reference ID/Investigator# 23162, Brussels
  - Site Reference ID/Investigator# 23843, Edegem
  - Site Reference ID/Investigator# 23161, Ghent
  - Site Reference ID/Investigator# 23842, Gilly
  - Site Reference ID/Investigator# 23163, Leuven
- Canada (6):
  - Site Reference ID/Investigator# 26702, Edmonton
  - Site Reference ID/Investigator# 25482, Halifax
  - Site Reference ID/Investigator# 39614, Montreal
  - Site Reference ID/Investigator# 23184, Ottawa
  - Site Reference ID/Investigator# 23183, Sherbrooke
  - Site Reference ID/Investigator# 24522, Toronto
- Chile (2):
  - Site Reference ID/Investigator# 36967, Temuco
  - Site Reference ID/Investigator# 36964, Viña del Mar
- China (17):
  - Site Reference ID/Investigator# 23186, Beijing
  - Site Reference ID/Investigator# 43443, Changchun
  - Site Reference ID/Investigator# 23194, Chengdu
  - Site Reference ID/Investigator# 43442, Chongqing
  - Site Reference ID/Investigator# 44444, Dalian
  - Site Reference ID/Investigator# 43444, Fuzhou
  - Site Reference ID/Investigator# 43482, Guangzhou
  - Site Reference ID/Investigator# 42563, Hangzhou
  - Site Reference ID/Investigator# 44443, Harbin
  - Site Reference ID/Investigator# 44062, Jinan
  - Site Reference ID/Investigator# 23191, Nanjing
  - Site Reference ID/Investigator# 44063, Nanning
  - Site Reference ID/Investigator# 42817, Qingdao
  - Site Reference ID/Investigator# 40624, Shanghai
  - Site Reference ID/Investigator# 23189, Shanghai
  - Site Reference ID/Investigator# 40448, Suzhou
  - Site Reference ID/Investigator# 23190, Xi'an
- Czechia (6):
  - Site Reference ID/Investigator# 23167, Brno
  - Site Reference ID/Investigator# 23166, Olomouc
  - Site Reference ID/Investigator# 24523, Prague
  - Site Reference ID/Investigator# 23844, Prague
  - Site Reference ID/Investigator# 40930, Prague
  - Site Reference ID/Investigator# 23197, Ústí nad Labem
- Site Reference ID/Investigator# 23442, Aarhus C, Denmark
- Egypt (2):
  - Site Reference ID/Investigator# 23198, Alexandria
  - Site Reference ID/Investigator# 23199, Cairo
- France (9):
  - Site Reference ID/Investigator# 43302, Amiens
  - Site Reference ID/Investigator# 23201, Clichy
  - Site Reference ID/Investigator# 43144, Créteil
  - Site Reference ID/Investigator# 23200, Lille
  - Site Reference ID/Investigator# 23168, Paris
  - Site Reference ID/Investigator# 40623, Paris
  - Site Reference ID/Investigator# 28345, Rouen
  - Site Reference ID/Investigator# 23165, Strasbourg
  - Site Reference ID/Investigator# 28347, Vandœuvre-lès-Nancy
- Germany (5):
  - Site Reference ID/Investigator# 23267, Berlin
  - Site Reference ID/Investigator# 23845, Bochum
  - Site Reference ID/Investigator# 23266, Frankfurt am Main
  - Site Reference ID/Investigator# 23268, Freiburg im Breisgau
  - Site Reference ID/Investigator# 23269, Mainz
- Site Reference ID/Investigator# 24525, Athens, Greece
- Site Reference ID/Investigator# 24980, Hong Kong, Hong Kong
- Italy (7):
  - Site Reference ID/Investigator# 27998, Benevento
  - Site Reference ID/Investigator# 23424, Milan
  - Site Reference ID/Investigator# 41488, Milan
  - Site Reference ID/Investigator# 23425, Palermo
  - Site Reference ID/Investigator# 41542, Pavia
  - Site Reference ID/Investigator# 23428, Rome
  - Site Reference ID/Investigator# 24042, Rome
- Japan (20):
  - Site Reference ID/Investigator# 26506, Aichi
  - Site Reference ID/Investigator# 36308, Chiba
  - Site Reference ID/Investigator# 37602, Chiba
  - Site Reference ID/Investigator# 29758, Fukuoka
  - Site Reference ID/Investigator# 37603, Hokkaido
  - Site Reference ID/Investigator# 28189, Ibaraki-ken
  - Site Reference ID/Investigator# 26505, Kanazawa
  - Site Reference ID/Investigator# 29757, Kumamoto
  - Site Reference ID/Investigator# 27343, Kurume
  - Site Reference ID/Investigator# 29759, Matsuyama
  - Site Reference ID/Investigator# 26507, Osaka
  - Site Reference ID/Investigator# 27959, Osaka
  - Site Reference ID/Investigator# 26508, Sayama
  - Site Reference ID/Investigator# 29756, Shimotsuke
  - Site Reference ID/Investigator# 36782, Shizuoka
  - Site Reference ID/Investigator# 28187, Tochigi-ken
  - Site Reference ID/Investigator# 26503, Tokyo
  - Site Reference ID/Investigator# 27242, Tokyo
  - Site Reference ID/Investigator# 26504, Yokohama
  - Site Reference ID/Investigator# 26509, Yufu
- Malaysia (3):
  - Site Reference ID/Investigator# 23461, George Town
  - Site Reference ID/Investigator# 23460, Kuala Lumpur
  - Site Reference ID/Investigator# 23459, Petaling Jaya, Selangor
- Mexico (3):
  - Site Reference ID/Investigator# 23155, Durango, DGO.
  - Site Reference ID/Investigator# 43102, Monterrey, NL
  - Site Reference ID/Investigator# 43145, Monterrey, NL
- Netherlands (3):
  - Site Reference ID/Investigator# 23272, Amsterdam
  - Site Reference ID/Investigator# 23270, Amsterdam
  - Site Reference ID/Investigator# 24782, Rotterdam
- Site Reference ID/Investigator# 23160, Auckland, New Zealand
- Site Reference ID/Investigator# 23846, Oslo, Norway
- Puerto Rico (2):
  - Site Reference ID/Investigator# 42706, Ponce
  - Site Reference ID/Investigator# 42705, San Juan
- Romania (6):
  - Site Reference ID/Investigator# 33979, Baia Mare
  - Site Reference ID/Investigator# 33344, Bucharest
  - Site Reference ID/Investigator# 33343, Cluj-Napoca
  - Site Reference ID/Investigator# 33977, Craiova
  - Site Reference ID/Investigator# 33345, Iași
  - Site Reference ID/Investigator# 33346, Oradea
- Russia (4):
  - Site Reference ID/Investigator# 43202, Chelyabinsk
  - Site Reference ID/Investigator# 43203, Kazan'
  - Site Reference ID/Investigator# 23462, Moscow
  - Site Reference ID/Investigator# 23849, Moscow
- Singapore (2):
  - Site Reference ID/Investigator# 23159, Singapore
  - Site Reference ID/Investigator# 23158, Singapore
- South Korea (12):
  - Site Reference ID/Investigator# 23447, Busan
  - Site Reference ID/Investigator# 39003, Busan
  - Site Reference ID/Investigator# 23445, Busan
  - Site Reference ID/Investigator# 23444, Daegu
  - Site Reference ID/Investigator# 26543, Gyeonggi-do
  - Site Reference ID/Investigator# 23457, Jeollanam-do
  - Site Reference ID/Investigator# 39002, Jeonju
  - Site Reference ID/Investigator# 23454, Seoul
  - Site Reference ID/Investigator# 25562, Seoul
  - Site Reference ID/Investigator# 23449, Seoul
  - Site Reference ID/Investigator# 23456, Seoul
  - Site Reference ID/Investigator# 23450, Suwon
- Spain (7):
  - Site Reference ID/Investigator# 23466, A Coruña
  - Site Reference ID/Investigator# 26063, Madrid
  - Site Reference ID/Investigator# 40931, Madrid
  - Site Reference ID/Investigator# 23465, Madrid
  - Site Reference ID/Investigator# 23463, Madrid
  - Site Reference ID/Investigator# 23467, Santander
  - Site Reference ID/Investigator# 23468, Zaragoza
- Taiwan (12):
  - Site Reference ID/Investigator# 23475, Changhua
  - Site Reference ID/Investigator# 23472, Kaohsiung County
  - Site Reference ID/Investigator# 25262, Taichung
  - Site Reference ID/Investigator# 23474, Taichung
  - Site Reference ID/Investigator# 23476, Tainan
  - Site Reference ID/Investigator# 23478, Tainan
  - Site Reference ID/Investigator# 23477, Tainan
  - Site Reference ID/Investigator# 23470, Taipei
  - Site Reference ID/Investigator# 43237, Taipei
  - Site Reference ID/Investigator# 23473, Taipei
  - Site Reference ID/Investigator# 23469, Taipei
  - Site Reference ID/Investigator# 23471, Taoyuan District

REFERENCES:
- [Derived] Kolamunnage-Dona R, Berhane S, Potts H, Williams EH, Tanner J, Janowitz T, Hoare M, Johnson P. Sorafenib is associated with a reduced rate of tumour growth and liver function deterioration in HCV-induced hepatocellular carcinoma. J Hepatol. 2021 Oct;75(4):879-887. doi: 10.1016/j.jhep.2021.05.015. Epub 2021 May 27. PMID 34052255
- [Derived] Cainap C, Qin S, Huang WT, Chung IJ, Pan H, Cheng Y, Kudo M, Kang YK, Chen PJ, Toh HC, Gorbunova V, Eskens FA, Qian J, McKee MD, Ricker JL, Carlson DM, El-Nowiem S. Linifanib versus Sorafenib in patients with advanced hepatocellular carcinoma: results of a randomized phase III trial. J Clin Oncol. 2015 Jan 10;33(2):172-9. doi: 10.1200/JCO.2013.54.3298. Epub 2014 Dec 8. PMID 25488963